CLINICAL TRIAL: NCT04308187
Title: The COVISTRESS Study: Influence of the COvid-19 Epidemic on STRESS
Brief Title: Influence of the COvid-19 Epidemic on STRESS
Acronym: COVISTRESS
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: University Hospital, Clermont-Ferrand (Other)
Collaborators: UMR CNRS 6024 LaPSCo, Clermont-Ferrand, France (Unknown); Wittyfit, Paris, France (Unknown)
Responsible Party: Sponsor
Other Study IDs: 2020 COVISTRESS
Record Dates: First submitted 2020-03-12; First posted 2020-03-13 (Actual); Last update posted 2020-03-13 (Actual); Status verified 2020-03

CONDITIONS: Stress, Psychological
Keywords: Stress, Psychological; Coronavirus; Epidemics
MeSH Terms: conditions — Stress, Psychological; Coronavirus Infections

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Patient Registry: Yes
Target Follow-Up Duration: 1 Day
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
The Coronavirus has a major influence on stress for the general population. However, data are currently non-existent concerning the perception and knowledge of the epidemic, the feeling of information from companies / establishments / governments, the means of protection used, the feelings of fear generated and their impact on feelings of stigmatization towards certain ethnic groups or categories of patients (those who cough ...), or relationships with socio-demographic factors or lifestyle.

DETAILED DESCRIPTION:
This is an observational study using a REDCap® questionnaire via an internet link, which will be distributed by any means (Facebook, Twitter, institution mailing lists via a referent, flash codes distributed to patients and the public, etc.).

The self-questionnaire will assess stress, perception and knowledge of the epidemic, the feeling of information on the part of businesses / establishments / governments, the means of protection used the feelings of fear generated and their impact on feelings of stigmatization towards certain ethnic groups or categories of patients (those who cough ...), or relationships with socio-demographic factors or lifestyle.

ELIGIBILITY:
Inclusion Criteria:

* Anyone volunteer to participate

Exclusion Criteria:

* Anyone non-voluntary to participate

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: General population
Sampling Method: Non-Probability Sample
Enrollment: 50000 (Estimated)
Dates: Start 2020-03-11 (Estimated); Primary Completion 2022-03 (Estimated); Study Completion 2022-03 (Estimated)

PRIMARY OUTCOMES:
Stress | Day 1
  Stress level will be assessed by questionnaire

SECONDARY OUTCOMES:
Perception and knowledge of the epidemic | Day 1
  Perception and knowledge of the epidemic will be assessed by questionnaire
Feeling of information on the part of companies / establishments / governments | Day 1
  The feeling of information will be assessed by questionnaire
Means of protection | Day 1
  the means of protection used will be assessed by questionnaire
Feelings of fear generated and its impact on feelings of stigmatization towards ethnic groups or categories of patients | Day 1
  The feeling of fear and the impact on stigmatization will be assessed by questionnaire
Sociodemographic factors and lifestyle habits | Day 1
  Sociodemographic factors and lifestyle habits will be assessed by questionnaire

CONTACTS AND LOCATIONS:
Overall Officials: Fréderic DUTHEIL, Principal Investigator — University Hospital, Clermont-Ferrand
Locations (1):
- University Hospital, Clermont-Ferrand, Clermont-Ferrand, France